CLINICAL TRIAL: NCT03402178
Title: A Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Studies to Assess the Safety, Tolerability, and Pharmacokinetics of E2082 in Healthy Male Subjects
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2082 in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety Review
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2082-J081-001
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Healthy Participants
Keywords: E2082; male; single ascending dose; multiple ascending dose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E2082 (Experimental): E2082 will be administered as a solution (0.2 milligram [mg]), a 0.5 mg tablet, and a 5 mg tablet. Part A: Cohort 1 participants will receive a single dose of a 0.2 mg E2082 solution, and participants in Cohorts 2 to 4, respectively, will receive a single dose of 0.5 mg, 1 mg, or 2.5 mg E2082 tablets under fasted conditions. Cohort 5 participants will receive a single dose of 5 mg E2082 under fasted conditions, and then they will receive 5 mg E2082 under fed conditions after washout. Participants in Cohorts 6 to 10, respectively, will receive 10 mg (adult participants), 15 mg, 25 mg, 40 mg, or 10 mg (elderly participants) E2082 tablets under fasted conditions. Part B: Participants in Cohorts 1 to 4, respectively, will receive 2.5 mg, 5 mg, 10, or 15 mg tablets once daily for 10 days. E2082 will be administered under fasted conditions on Day 1 and Day 10 and under fed conditions during Day 2 to Day 9.
  Interventions: Drug: E2082
- E2082-matched placebo (Placebo Comparator): Matched placebo will be administered as a solution (0.2 mg), a 0.5 mg tablet, and a 5 mg tablet. Part A: Cohort 1 participants will receive a single dose of a 0.2 mg matched placebo solution, and participants in Cohorts 2 to 4, respectively, will receive a single dose of 0.5 mg, 1 mg, or 2.5 mg matched placebo tablets under fasted conditions. Cohort 5 participants will receive a single dose of 5 mg matched placebo under fasted conditions, and then they will receive 5 mg matched placebo under fed conditions after washout. Participants in Cohorts 6 to 10, respectively, will receive 10 mg (adult participants), 15 mg, 25 mg, 40 mg, or 10 mg (elderly participants) matched placebo tablets under fasted conditions. Part B: Participants in Cohorts 1 to 4, respectively, will receive 2.5 mg, 5 mg, 10, or 15 mg matched placebo tablets once daily for 10 days. Matched placebo will be administered under fasted conditions on Day 1 and Day 10 and under fed conditions during Day 2 to Day 9.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2082 — Solution (0.2 mg) or tablet (0.5 mg and 5 mg).
  Arms: E2082
Drug: Placebo — Solution (0.2 mg) or tablet (0.5 mg and 5 mg) matched to E2082.
  Arms: E2082-matched placebo

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, and pharmacokinetics (PK) of single ascending oral doses of E2082 in healthy Japanese adult and elderly male participants, and to evaluate the safety, tolerability, and PK of multiple ascending oral doses of E2082 in healthy Japanese and Caucasian adult male participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

* Non-smoking, age ≥20 years and <55 years old adult male (Cohorts 1 to 9 of Part A and all cohorts of Part B), or age ≥55 years and ≤85 years old elderly male (only Cohort 10 of Part A) at the time of informed consent. To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing.
* Body mass index ≥18 and <30 kilograms per meters squared at Screening

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

* Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
* Any history of gastrointestinal surgery that may affect pharmacokinetic profiles of E2082, example, hepatectomy, nephrectomy, and digestive organ resection
* Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram finding, or laboratory test results that require medical treatment at Screening

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Part A: Mean value of the maximum observed concentration (Cmax) of E2082 under a fasted state for the single ascending dose (SAD) Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  Cmax is the maximum observed concentration of E2082 in the plasma that is measured after a dose.
Part A: Mean value of Cmax of E2082 under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  Cmax is the maximum observed concentration of E2082 in the plasma that is measured after a dose.
Part A: Mean value of the time at which the highest plasma concentration (Tmax) of E2082 occurs under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  Tmax is the time at which the highest concentration of E2082 occurs.
Part A: Mean value of Tmax of E2082 under fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  Tmax is the time at which the highest concentration of E2082 occurs.
Part A: Mean value of the area under the concentration-time curve from zero time to 24 hours after dosing (AUC[0-24h]) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
  AUC(0-24h) represents the total drug exposure from zero time to 24 hours after dosing.
Part A: Mean value of AUC(0-24h) under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose
  AUC(0-24h) represents the total drug exposure from zero time to 24 hours after dosing.
Part A: Mean value of AUC from zero time to the time of the last quantifiable concentration (AUC[0-t]) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  AUC(0-t) represents the total drug exposure from zero time to the time of the last quantifiable concentration.
Part A: Mean value of AUC(0-t) under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  AUC(0-t) represents the total drug exposure from zero time to the time of the last quantifiable concentration.
Part A: Mean value of AUC from zero time to 72 hours after dosing (AUC[0-72h]) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours postdose
  AUC(0-72h) represents the total drug exposure from zero time to 72 hours after dosing.
Part A: Mean value of AUC(0-72h) under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hours postdose
  AUC(0-72h) represents the total drug exposure from zero time to 72 hours after dosing.
Part A: Mean value of AUC from zero time to 96 hours after dosing (AUC[0-96h]) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours postdose
  AUC(0-96h) represents the total drug exposure from zero time to 96 hours after dosing.
Part A: Mean value of AUC(0-96h) under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours postdose
  AUC(0-96h) represents the total drug exposure from zero time to 96 hours after dosing.
Part A: Mean value of AUC from zero time extrapolated to infinite time (AUC[0-inf]) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  AUC(0-inf) represents the total drug exposure from zero time extrapolated to infinite time.
Part A: Mean value of AUC(0-inf) under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  AUC(0-inf) represents the total drug exposure from zero time extrapolated to infinite time.
Part A: Mean value of terminal elimination phase half-life (t½) of E2082 under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  t½ is the time required for the concentration or amount of drug in the body to be reduced to exactly one-half of a given concentration or amount.
Part A: Mean value of t½ of E2082 under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  t½ is the time required for the concentration or amount of drug in the body to be reduced to exactly one-half of a given concentration or amount.
Part A: Mean value of apparent total clearance (CL/F) of E2082 under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), and 168 (Day 8) hours postdose for all cohorts. Additionally, 240 (Day 11) and 336 (Day 15) hours postdose for Cohort 4 or later.
  CL/F is the apparent total clearance following extravascular (example, oral) administration.
Part A: Mean value of CL/F of E2082 under a fasted state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 168 (Day 8), 240 (Day 11), and 336 (Day 15) hours postdose
  CL/F is the apparent total clearance following extravascular (example, oral) administration.
Part A: Mean value of the apparent volume of distribution at terminal phase of E2082 on Day 1 (Vz/F) under a fasted state for the SAD Cohorts 1-10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 12 hours postdose
  The apparent volume of distribution gives information about the amount of drug distributed in body tissue rather than the plasma.
Part A: Mean value of Vz/F of E2082 on Day 1 under a fed state for the SAD Cohort 5 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 12 hours postdose
  The apparent volume of distribution gives information about the amount of drug distributed in body tissue rather than the plasma.
Part B: Mean value of Cmax of E2082 for the multiple ascending dose (MAD) cohorts on Day 1 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1
  Cmax is the maximum observed concentration of E2082 in the plasma that is measured after a dose.
Part B: Mean value of Cmax of E2082 at steady state (Css,max) for the MAD cohorts on Day 10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  Cmax is the maximum observed concentration of E2082 in the plasma that is measured after a dose.
Part B: Mean value of the minimum observed concentration (Cmin) of E2082 for the MAD cohorts on Day 1 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1
  Cmin is the minimum observed concentration of E2082 in the plasma that is measured after a dose.
Part B: Mean value of Cmin of E2082 at steady state (Css,min) for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  Css,min is the minimum observed concentration of E2082 in the plasma that is measured after a dose at steady state.
Part B: Mean value of Tmax of E2082 for the MAD cohorts on Day 1 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1
  Tmax is the time at which the highest concentration of E2082 occurs.
Part B: Mean value of Tmax of E2082 at steady state (Tss,max) for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  Tss,max is the time at which the highest concentration of E2082 occurs at steady state.
Part B: Mean value of the average steady state concentration (Css,av) of E2082 for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 10
  The average steady state concentration is calculated as AUC(0-τ)/τ. τ is the dosing interval.
Part B: Mean value of AUC(0-24h) after dosing on Day 1 for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1
  AUC(0-24h) represents the total drug exposure from zero time to 24 hours after dosing.
Part B: Mean value of AUC(0-τ) for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose of Day 10
  AUC(0-τ) is AUC over the dosing interval on multiple dosing.
Part B: Mean value of t½ following the last day of dosing for the MAD cohorts | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  t½ is the time required for the concentration or amount of drug in the body to be reduced to exactly one-half of a given concentration or amount.
Part B: Peak-trough fluctuation (PTF) for the MAD cohorts | Predose at Days 1, 2, 6, 10, 12, 13, and 14. 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1. 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  PTF is peak to trough fluctuation at steady-state.
Part B: Accumulation ratio for AUC and Cmax (Rac) for the MAD cohorts | Predose at Days 1, 2, 6, 10, 12, 13, and 14. 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose of Day 1. 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  Rac (Cmax) is calculated as the ratio of drug concentrations observed during a dosing interval at steady-state divided by drug concentrations seen during the dosing interval after a single (first) dose. Rac (AUC)=steady state AUC(0-τ)/single dose AUC(0- τ), where τ is dosing interval.
Part B: Mean value of apparent total clearance at steady state (CLss/F) for the MAD cohorts on Day 10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  CLss/F is the apparent total clearance at steady state following extravascular (example, oral) administration. It is defined as the rate of drug elimination.
Part B: Mean value of Vz/F for the MAD cohorts on Day 10 | Predose and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 168, 240, and 336 hours postdose of Day 10
  Vz/F is apparent volume of distribution at terminal phase on Day 10.
Part B: Change from baseline in QT interval corrected for heart rate using the Fridericia formula (QTcF) | Baseline and Day 1
Part B: Change from baseline in QT interval corrected for heart rate using the Fridericia formula (QTcF) | Baseline and Day 10

SECONDARY OUTCOMES:
Change-from-baseline in heart rate (HR) | Baseline, Days 1 and 10
Change from baseline in PR interval and QRS interval of the Electrocardiogram (ECG) | Baseline, Days 1 and 10
Placebo-corrected change from baseline in HR | Baseline, Days 1 and 10
Placebo-corrected change from baseline in QTcF, PR, QRS interval | Baseline, Days 1 and 10
Number of participants with categorical outliers for HR, PR interval, QRS interval | Baseline up to Day 11
Number of participants with categorical outliers defined as QTcF >450 msec, 480 msec and 500 msec at any timepoint and change-from-baseline QTcF (ΔQTcF) >30 msec (increased by 30 msec) and >60 msec | Baseline up to Day 11
Number of participants with T wave morphology changes | Baseline up to Day 11
Number of participants with U-wave presence | Baseline up to Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site, Sumida-ku, Tokyo, Japan